CLINICAL TRIAL: NCT00807326
Title: A Randomized, Parallel Group Comparison of Loperamide/Simeticone Caplet, Loperamide/Simeticone Chewable Tablet (IMODIUM® PLUS) and a Probiotic (Saccharomyces Boulardii) in the Treatment of Acute Diarrhea in Adults
Brief Title: A Comparison of Three Medications to Treat Diarrhea in Adults.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOPDIR4002
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Diarrhea
Keywords: Antidiarrheals
MeSH Terms: conditions — Diarrhea | interventions — Loperamide; Simethicone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Loperamide/simeticone Caplets (Experimental): Drug (including placebo)
  Interventions: Drug: Loperamide/simeticone 2 mg/125 mg caplets
- Loperamide/simeticone Chewable Tablets (Active Comparator): Drug (including placebo)
  Interventions: Drug: Loperamide/simeticone 2 mg/125 mg chewable tablets
- Probiotic Capsules (Active Comparator): Drug (including placebo)
  Interventions: Drug: Probiotic Saccharomyces boulardii 250 mg capsules

INTERVENTIONS:
Drug: Loperamide/simeticone 2 mg/125 mg caplets — Oral, 2 caplets taken initially at investigator site followed by one caplet after each unformed stool, maximum 4 caplets in a 24 hour period for a maximum of 48 hours (per product label)
  Other Names: Imodium® Plus Caplet
  Arms: Loperamide/simeticone Caplets
Drug: Loperamide/simeticone 2 mg/125 mg chewable tablets — Oral, 2 chewable tablets taken initially at the site followed by one chewable tablet after each unformed stool, maximum 4 chewable tablets in a 24 hour period for a maximum of 48 hours (per product label)
  Other Names: Imodium® Plus Chewable tablet
  Arms: Loperamide/simeticone Chewable Tablets
Drug: Probiotic Saccharomyces boulardii 250 mg capsules — Oral, 1 capsule twice a day, maximum 2 capsules in a 24 hour period for a maximum of 5 days (per product label)
  Other Names: Perenterol® Forte 250mg capsules
  Arms: Probiotic Capsules

SUMMARY:
A comparison of three medications to treat diarrhea in adults.

DETAILED DESCRIPTION:
This single (investigator) blind, randomized, 3-arm, parallel-group study design was selected to show non-inferiority of loperamide/simeticone caplets compared to chewable tablets in a heterogeneous subject population aiming at validity of results and reducing bias. The study will also compare the loperamide/simeticone combinations versus a probiotic (Saccharomyces boulardii) in the treatment of acute diarrhea in adults. Probiotics have been used for acute infectious diarrhea to reduce the duration and severity of the illness.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age
* Acute diarrhea illness with symptoms onset within 48 hours of study entry
* Minimum of 3 unformed stools in 24 hours before study entry
* Most recent stool is unformed
* Abdominal discomfort/wind (intensity mild to severe) within 4 hours of study entry
* Women of childbearing potential must have a negative pregnancy test at screening
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Requiring hospital admission, parenteral hydration or antibiotic therapy Axillary temperature >38.2°C or oral temperature >38.6°C
* History or clinical evidence of gross blood or pus in stool in current illness
* Signs or symptoms of orthostatic hypotension
* Unable to take medication and fluids by mouth
* History of chronic gastrointestinal disease, hepatic or renal insufficiency, or other significant medical condition that could be aggravated by untreated acute diarrhea
* Immunodeficiency (e.g. those with acquired immunodeficiency syndrome [AIDS] or known human immunodeficiency virus [HIV] infection, or undergoing chemotherapy or radiotherapy)
* Intake of antibiotics, oral antifungals, quinidine or ritonavir within 7 days, antidiarrhoeal, promotility drugs (e.g., metoclopramide, domperidone), antiflatulents (e.g., simeticone, activated charcoal) or probiotics or bismuth salts within 48 hours, or any analgesic within 6 hours prior to study entry Hypersensitivity to loperamide, yeast, or any component of study formulations
* Pregnant or breast-feeding
* Unable to comply with the protocol requirements and schedule
* Any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study
* Use of opiates (as 'recreational' drugs and as painkillers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Number of unformed stools | 0-24 hours

SECONDARY OUTCOMES:
Number of unformed stools | 0-12, 12-24, 24-36, 36-48 hours
Time to last unformed stool | Throughout duration of the study
Time to complete relief of abdominal discomfort | Throughout duration of the study
Time to complete relief of diarrhea | Throughout duration of the study
Proportion of subjects with complete relief of diarrhea | 4, 8, 12, 24 and 48 hours
Gas-related abdominal discomfort ratings - change from baseline at subsequent time points | Throughout duration of the study
Proportions of subjects with complete well-being | at 12, 24 and 48 hours.
Subject's evaluation of treatment effectiveness for overall illness relief, diarrhea relief and abdominal discomfort relief | Throughout duration of the study
Number of loperamide/simeticone 2 mg/125 mg caplets or chewable tablets or probiotic (Saccharomyces boulardii) 250 mg capsules used during the study | Throughout duration of the study
Frequency of complete well-being following diarrhea illness | at 7 days follow up
Stool frequency | at 7 days follow up
Frequency of diarrhea relapse | at 7 days follow up
Safety Assessments will consist of monitoring and recording all non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs), their frequency, severity, seriousness, and relationship to the investigational product. | throughout duration of the study (+ 30 days for spontaneously-reported SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (6):
- India (2):
  - Manipal Goa Hospital, Mormugao, Goa
  - Vrundavan Hospital & Research Centre, Mormugao, Goa
- Mexico (4):
  - North West Medical, San José del Cabo, Baja California Sur
  - Dr. Maxwell´s Clinic, San Miguel de Allende, Guanuajuato
  - Hospital Amerimed Puerto Vallarta, Puerto Vallarta, Jalisco
  - Servicios Medicos de la Bahia, Puerto Vallarta, Jalisco

REFERENCES:
- [Derived] Cottrell J, Koenig K, Perfekt R, Hofmann R; Loperamide-Simethicone Acute Diarrhoea Study Team. Comparison of Two Forms of Loperamide-Simeticone and a Probiotic Yeast (Saccharomyces boulardii) in the Treatment of Acute Diarrhoea in Adults: A Randomised Non-Inferiority Clinical Trial. Drugs R D. 2015 Dec;15(4):363-73. doi: 10.1007/s40268-015-0111-y. PMID 26541878